CLINICAL TRIAL: NCT01225406
Title: Treatment Cohort of HIV-infected Children With Resistance or Intolerance to Non Nucleoside Reverse Transcriptase Inhibitor (NNRTI) First Line and PI Second Line Antiretroviral Therapy
Brief Title: Third Line Highly Active Antiretroviral Therapy (HAART) in HIV-infected Children
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Ministry of Education, Thailand (Other); National Health Security Office, Thailand (Other)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 113
Record Dates: First submitted 2010-10-18; First posted 2010-10-21 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: This Study is Designed to Collect Treatment Data of Thai Children on Third Line ARV Therapy
Keywords: Third line ARV therapy; HIV RNA; Absolute CD4+ T cell count; serious adverse events (SAEs); Drug resistance
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Plasma and PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- third line naive: Children on second line or other regimen who switch or start third line regimen
  Interventions: Drug: Tenofovir
- third line experienced: children who are on third line regimen
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir

SUMMARY:
This is an observational cohort study of virologic and immunologic outcome after at least 48 weeks of third line antiretroviral therapy. Upto 150 children at 8 Thai sites will be enrolled. Third line antiretroviral therapy in this study is defined as an antiretroviral (ARV) regimen in a patient who has failure or intolerance to first line NNRTI-based therapy and second line PI-based therapy. Such regimens may contain new drugs or drug classes such as darunavir, tipranavir, etravirine and raltegravir The knowledge gained from this study will help the Thai government in planning its strategy to provide third line ARV therapy to children within the national program.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the virological efficacy, as measured by the proportions of children with HIV RNA below 400 and 50 copies/ml at 48 weeks after initiating third line ARV therapy.

Third line ARV therapy is defined as an ARV regimen in a patient who has failure or intolerance to first line NNRTI-based therapy and second line PI-based therapy. Such regimens may contain new drugs or drug classes such as darunavir, tipranavir, etravirine and raltegravir

ELIGIBILITY:
Inclusion Criteria:

Children (< 18 years old) with HIV infection may enroll if one of the following criteria is met:

1. Have resistance to at least one drug in each of the 3 classes (NRTI, NNRTI and PI) and have plasma HIV RNA > 1000 copies/ml prior to switching to third line ARV therapy
2. Have intolerance to the current NRTI, NNRTI or PI treatment and need to receive darunavir, etravirine, tipranavir or raltegravir

Exclusion Criteria:

1. Have hepatic impairment with ALT ≥ 5 upper limit of normal
2. Pregnant or breastfeeding

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Thai children aged < 18 years old who are on or are switching to third line antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
undetectable viral load | 48 weeks
  Primary endpoint will be the proportions of subjects with HIV RNA below 400 and 50 copies/ml at 48 weeks.

SECONDARY OUTCOMES:
Hyperlipidemia | 48 weeks
  Number of subjects with hyperlipidemia as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Thanyawee Puthanakit, MD, Principal Investigator — Chulalongkorn University Bangkok; Kulkanya Chokephaibulkit, MD, Principal Investigator — Siriraj Hospital
Locations (9):
- Thailand (9):
  - Prapokklao Chantaburi, Chanthaburi, Changwat Chanthaburi
  - Chulalongkorn University, Bangkok
  - HIV-NAT, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
  - Nakornping Hospital, Chiang Mai
  - Chiang Rai Regional Hospital, Chiang Rai
  - Khon Kaen University, Khon Kaen
  - Bamrasnaradura Institute, Nonthaburi
  - Surin Hospital, Surin

REFERENCES:
- [Result] Chokephaibulkit K, Prasitsuebsai W, Wittawatmongkol O, Gorowara M, Phongsamart W, Sophonphan J, Kerr SJ, Vanprapar N, Puthanakit T, Pasomsap C, Suwanlerk T, Sekar V, Burger D, Ananworanich J; HIV-NAT 113 Pharmacokinetic Study Group. Pharmacokinetics of darunavir/ritonavir in Asian HIV-1-infected children aged >/=7 years. Antivir Ther. 2012;17(7):1263-9. doi: 10.3851/IMP2347. Epub 2012 Sep 6. PMID 22954687
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org